CLINICAL TRIAL: NCT02849613
Title: Regenerative Stem Cell Therapy for Stroke in Europe
Acronym: RESSTORE
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Not authorized by Regulatory agencies - new protocol phase 1a in progress
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Horizon 2020 - European Commission (Other); University Grenoble Alps (Other); Servicio Madrileño de Salud, Madrid, Spain (Other); St. Anne's University Hospital Brno, Czech Republic (Other); Andaluz Health Service (Other Government); University of Glasgow (Other); University of Eastern Finland (Other); Etablissement Français du Sang (Other); Tampere University (Other); Histocell SL, Spain (Unknown); Oy Medfiles Ltd (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Hospices Civils de Lyon (Other); Association Groupe ESSEC (Other); NOVADISCOVERY SAS, France (Unknown); Finovatis (Other); Centre Hospitalier Universitaire de Besancon (Other); Assistance Publique - Hôpitaux de Paris (Other); University Hospital, Toulouse (Other); University Hospital, Bordeaux (Other); University Hospital, Caen (Other); Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Servicio de Salud de Castilla La Mancha, Albacete, Spain (Unknown); Servicio Gallego de Salud (Other Government); Pirkanmaa Hospital District, Tampere, Finland (Unknown); Hospital Vall d'Hebron (Other); Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 38RC15.337
Record Dates: First submitted 2016-07-06; First posted 2016-07-29 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2016-07

CONDITIONS: Stroke
Keywords: cell therapy; stem cell; transplantation; graft; recovery; repair; stroke; mesenchymal stem cell; regenerative
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adipose derived Stem Cells ADSC (Experimental): ADSC, single IV, 1.106 cells/kg
  Interventions: Other: Adipose Derived Stem Cells
- Vehicle media (Sham Comparator): IV infusion of cell excipients, 1ml/kg
  Interventions: Other: Vehicle media

INTERVENTIONS:
Other: Adipose Derived Stem Cells
  Other Names: ADSC
  Arms: Adipose derived Stem Cells ADSC
Other: Vehicle media
  Other Names: Placebo
  Arms: Vehicle media

SUMMARY:
Stroke is the second leading cause of death in the world population. When not fatal, stroke often results in disability, and secondary health problems affecting not only patients but also their families. Building on emerging preclinical and pilot clinical evidences, RESSTORE will focus on the clinical assessment of regenerative cell therapy to improve stroke recovery and patients quality of life.

DETAILED DESCRIPTION:
RESSTORE European multicentre randomised phase IIb will explore the efficacy (functional recovery) and safety of intravenous infusion of allogenic adipose tissue derived mesenchymal stem cells (ADSC) in 400 stroke patients. Therapeutic effects of ADSCs will be assessed and monitored in patients using clinical rating scales, multimodal MRI and blood biomarkers.

The European regenerative therapy capacities (France, Spain, Finland, United Kingdom and Czech Republic), developed in RESSTORE will cover the full value chain in the field (large scale GMP cell production, clinical testing, biomarkers discovery, understanding of the restoring mechanisms, biobanking...).

ELIGIBILITY:
Inclusion Criteria:

* Hemispheric ischemic stroke (>1.5cm)
* Inclusion from 1 to 4 days post-stroke
* NIHSS > or = 7
* No craniectomy
* Able to follow a rehabilitation program
* Modified Rankin scale = 0 before stroke onset

Exclusion Criteria:

* Coma
* Severe leucoariosis
* Previous stroke
* Active endocarditis, pneumonia, AIDS, active hepatic disease due to HBV or HCV
* History of cancer
* Pregnancy, breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Between-group difference of NIHSS (stroke severity score) | 6 months after stroke onset

CONTACTS AND LOCATIONS:
Overall Officials: Olivier DETANTE, MD PhD, Principal Investigator — University Hospital Grenoble-Alpes, France; Exuperio DIEZ TEJEDOR, MD PhD, Principal Investigator — La Paz University Hospital, Madrid, Spain
Locations (1):
- University Grenoble Hospital / EFS, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided